CLINICAL TRIAL: NCT02994563
Title: Amnis Therapeutics Thrombectomy Device-First in Man (FIM) Safety and Performance Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Subject recruitment problem due to Covid pandemic
Sponsor: Amnis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AmGR01
Record Dates: First submitted 2016-12-05; First posted 2016-12-16 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open arm (Experimental): Thrombectomy device to be used to retrieve clot and restore blood flow.
  Interventions: Device: Thrombectomy Device

INTERVENTIONS:
Device: Thrombectomy Device — The Amnis Thrombectomy Device is intended to restore blood flow by removing thrombus from intracranial vessels in patients experiencing ischemic stroke

SUMMARY:
Prospective, single-arm, open label, Safety and Performance clinical investigation.

DETAILED DESCRIPTION:
The Amnis Thrombectomy Device is intended to restore blood flow by removing thrombus from intracranial vessels in patients experiencing ischemic stroke. Pre-CE mark clinical investigation. Population will be subjects with documented untreated, acute ischemic stroke with large vessel occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Aged18-85years.
2. Subject who is contraindicated or failed (when the physician withdraws the tPA per physician discretion) intravenous tissue plasminogen activator (t-PA) therapy given at local institutions or within national practice. Failed means that the physician does not continue with IV tPA after thrombolysis; there is still an occlusion with TICI that is </= 1 as the relevant inclusion criteria.
3. Subject is able to be treated within 8 hours of stroke symptoms onset with minimum of one deployment of the Amnis Thrombectomy Device.
4. NIHSS score ≥8.
5. Pre-stroke mRS (modified Rankin Scale) score of 0 to 1.
6. Thrombolysis in cerebral infarction (TICI) ≤1 and causative occlusion of the M1 or M2 portion of the MCAs, anterior cerebral arteries, vertebral arteries, basilar artery ,or posterior cerebral arteries (P1 o rP2), confirmed by CT or MR angiography that is accessible to the Amnis thrombectomy device (i.e. according to IFU; 2-5.5 mm).
7. ASPECTS of ≥6 based on CT or MRI that was performed within 60 min prior to the start of endovascular procedure.
8. Subject or subject's legal guardian where regulations permit, signs the Patient Informed Consent and agrees that subject will attend follow-up visits.

Exclusion Criteria:

1. Rapid neurological improvement prior to or at time of treatment suggesting resolution of signs/symptoms of stroke.
2. Estimated time of symptom onset.
3. Baseline NIHSS score <8.
4. BaselineNIHSS score ≥30 or state of coma.
5. Baseline pre-stroke mRS score >1.
6. Baseline Thrombolysis in cerebral infarction (TICI) > 2a.
7. Known serious sensitivity to radiographic contrast agent.
8. Arterial tortuosity, pre-existing stent and/o rother arterial disease that would prevent the device from reaching the target vessel.
9. Evidence of a moderate/large core defined as extensive early ischemic changes of Alberta Stroke Program Early CT score (ASPECTS) <6.

   Co-morbid conditions:
10. Elevated blood pressure(systolic>185 mm Hg or diastolic >110 mm Hg)
11. Use of warfarin anticoagulation with INR >3.0.
12. Platelet count <30,000/mm³.
13. Blood glucose concentration <50 mg/dL (2.7 mmol/L).
14. CT/MRI imaging demonstrate smultilobar infarction (hypodensity >1/3 cerebral hemisphere).
15. CT or MRI evidence of mass effect, signs of hemorrhage, arteriovenous malformation or aneurysm or intra-cranial tumor (except small meningioma).
16. Angiographic evidence of carotid dissection, complete cervical carotid occlusions or vasculitis.
17. Clinical Symptoms or CT/MRI imaging suggest subarachnoid hemorrhage.
18. Imaging evidence that suggests, in the opinion of the investigator, the subject is not appropriate for mechanical thrombectomy intervention (e.g. inability to navigate to target lesion, moderate/large infarct with poor collateral circulation, etc.).

    General - related to the protocol or device:
19. Known sensitivity to nickel, titanium metals or their alloys.
20. Subject who requires hemodialysis or peritoneal dialysis, or who has a contraindication to an angiogram for whatever reason.
21. Current participation in another investigational drug or device study.
22. Female who is pregnant or lactating or has a positive pregnancy test at time of admission.
23. Subject currently uses or has a recent history of illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than four alcoholic drinks per day).
24. Subject has a life expectancy of <90 days.
25. Subject with a comorbid disease or condition that would confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
All serious adverse events (notably at 24 hours ± 3 hrs post procedure or until alternative stroke treatment is initiated, whichever comes first). | 24 hours ± 3 hrs post procedure or until alternative stroke treatment is initiated, whichever comes first.
  It will investigate whether the application of Amnis Thrombectomy device is a safe method, in acute stroke therapy, for obtaining recanalization of large vessels and with favorable patient outcome.
All cause mortality (90 days). | 3 months post-procedure
  Determine the number of participants with treatment-related adverse events.

SECONDARY OUTCOMES:
Arterial recanalization of the occluded target vessel in the immediate post-procedure angiogram. | Immediate post-procedure angiogram.
  Arterial recanalization of the occluded target vessel as angiographically scored by a Thrombolysis in Cerebral Infarction (TICI) flow grade of 2b or greater in the immediate post-procedure angiogram.
Proportion of patients with rapid neurological improvement as determined by a NIHSS ≤4. | First 24 hours after treatment
  Proportion of patients with rapid neurological improvement (more than 4 points on the NIHSS or NIHSS ≤4) during the first 24 hours after treatment.
Good functional clinical outcome as determine by a modified Rankin Scale score of 0-2. | First 24 hours after treatment.
  Proportion of patients with rapid neurological improvement (more than 4 points on the NIHSS or NIHSS ≤4) during the first 24 hours after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Andersson, M.D.; Ph.D., Principal Investigator — Karolinska Institute, Neuroradiology Clinic, Stockholm, Sweden
Locations (4):
- Spain (3):
  - Hospital Vall d'Hebron; Unidad Ictus, Barcelona
  - Hospital Clinico of Barcelona; Section of Vascular Radiology & Neuroradiology, Barcelona
  - Hospital Clínico Universitario (Valladolid); Dept. Neurology, Valladolid
- Karolinska Universitetssjukhuset i Solna, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No